CLINICAL TRIAL: NCT01216943
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Twice-daily 0.01% Bimatoprost/0.15% Brimonidine/0.5% Timolol Ophthalmic Solution (Triple Combination) in Patients in India, Who Have Glaucoma or Ocular Hypertension With Elevated IOP, and Are on Twice-daily 0.2% Brimonidine/0.5% Timolol Ophthalmic Solution (Dual Combination) Therapy
Brief Title: Safety and Efficacy of Triple Combination Therapy in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192024-049
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-07

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple Combination Therapy (Experimental): One drop of Triple Combination Therapy (bimatoprost/brimonidine tartrate/timolol fixed combination ophthalmic solution) administered to each eye, twice daily for 12 weeks.
  Interventions: Drug: bimatoprost/brimonidine tartrate/timolol fixed combination ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost/brimonidine tartrate/timolol fixed combination ophthalmic solution — One drop of Triple Combination Therapy (bimatoprost/brimonidine tartrate/timolol fixed combination ophthalmic solution) administered to each eye, twice daily for 12 weeks.

SUMMARY:
This study will investigate the safety and efficacy of Triple Combination Therapy (bimatoprost/brimonidine tartrate/timolol fixed combination ophthalmic solution) in patients with glaucoma or ocular hypertension who have elevated intraocular pressure (IOP) on brimonidine/timolol ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma and/or ocular hypertension in both eyes
* Requires IOP-lowering treatment in both eyes

Exclusion Criteria:

* Other active ocular disease other than glaucoma or ocular hypertension (eg, uveitis, ocular infections or severe dry eye)
* Current or anticipated use of ocular medications other than study medications, except for intermittent use of artificial tears
* Use of oral, injectable or topical corticosteroids within 21 days
* Iridectomy or laser peripheral iridotomy in the study eye within 3 months
* Uncomplicated cataract surgery in the study eye within 6 months
* Incisional glaucoma surgery in the study eye within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Coimbatore, Tamil Nadu, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triple Combination Therapy
Started | 126
Completed | 113
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 126
Age, Customized [Number; unit: Participants]
  <45 years | 11
  45 to 65 years | 84
  >65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the eye. Mean diurnal IOP is the mean of the IOP values at hour 0, hour 2 and hour 8 at each visit in the study eye. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase in IOP (worsening).
Time Frame: Baseline, Week 12
Population: Modified Intent to Treat: includes all qualified patients with a baseline and at least 1 postbaseline efficacy evaluation
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Triple Combination Therapy
Number analyzed (Participants) | 121
Millimeters of Mercury (mmHg)
  Baseline | 22.35 (3.417)
  Change from Baseline at Week 12 | -3.98 (2.856)

ADVERSE EVENTS:
Description: The Safety Population was used for adverse events (AEs) and serious adverse events (SAEs) and included all qualified treated patients.
Arm/Group | Triple Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/121
Other Adverse Events (participants affected / at risk) | 20/121
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=121)
Conjunctival Hyperaemia (Eye disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.